CLINICAL TRIAL: NCT05636202
Title: The Early Predictive Roles of NLR and NE% in In-hospital Mortality of Septic Patients: a Single-center 13-year Retrospective Study
Brief Title: The Role of NLR in the Diagnosis and Prognosis of Sepsis
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: NLR01
Record Dates: First submitted 2022-11-08; First posted 2022-12-05 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2022-10

CONDITIONS: Sepsis; Infections
Keywords: sepsis; NLR; Percentage of neutrophils; Prognosis
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survival group: Patients who survived sepsis
  Interventions: Other: No intervention
- Death group: Patients who died of sepsis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention in the retrospective study

SUMMARY:
Neutrophil-lymphocyte ratio (NLR), as an inflammatory index, is cheap and easy to obtain, and could be widely used in hospitals at all levels. NLR is a valuable biomarker that is significantly correlated with the status of immune and inflammatory responses. In the past few years, NLR has been continuously and extensively explored in various diseases, and the research progress is considerable. In cardiovascular disease, NLR can predict arrhythmia and short - and long-term mortality in patients with acute coronary syndrome. NLR may be associated with heart failure and valvular heart disease. Moreover, NLR has been shown to be associated with respiratory diseases (such as chronic obstructive pulmonary disease), immune diseases (rheumatoid arthritis and systemic lupus erythematosus), and digestive diseases (acute appendicitis, hepatocellular carcinoma, liver fibrosis, and cirrhosis).

Importantly, the study of NLR in sepsis has received much attention in recent years. A 2019 meta-analysis concluded that peripheral white blood cell ratios, including NLR, lymphocyte-to-monocyte ratio (LMR), and platelet-to-lymphocyte ratio (PLR), are associated with clinical outcomes in sepsis and are useful biomarkers of infection. They recommended that NLR be evaluated in future hierarchical models, To clarify its relationship with NLR and clinical outcome and the prognostic value of NLR, it is worth mentioning that NLR has also been found to have the ability to predict the outcome of sepsis. It has been shown that NLR, together with other inflammatory parameters, might be a marker for early detection of sepsis in the intensive care unit. However, a large body of evidence demonstrating the association between NLR and adverse clinical outcomes in sepsis remains controversial. Another study concluded that "no association was found between NLR and 28-day in-hospital mortality in patients with sepsis". In addition, the reliability of NLR on admission in predicting the prognosis of critical illness was also lower than that of traditional markers (including CRP, PCT, serum lactic acid and APACHEⅡ score).

This study aimed to retrospectively investigate the early predictive value of inflammation-related parameters in-hospital mortality of septic patients.

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening organ dysfunction caused by the host's malfunctioning response to infection, which has become one of the major problems in the world's public health. The development of effective biomarkers for the diagnosis of sepsis is undoubtedly helpful for us to timely and accurately understand the diagnosis, progression, and prognosis of sepsis.

The neutrophil-to-lymphocyte ratio (NLR), as an inflammatory indicator, is inexpensive and easily accessible parameter and could be widely used. In severe infectious diseases, particularly in sepsis, a substantial increase in peripheral blood neutrophils has been discovered, which reflects the severity of the inflammatory response. Neutrophil reverse migration following the initial neutrophil infiltration into inflammatory scenarios may further exacerbate the increase in the peripheral blood neutrophils. Lymphocyte apoptosis-induced reduction of peripheral blood lymphocytes is a significant feature of sepsis that could lead to adaptive immunosuppression. NLR is a cheap and rapidly available predictor of sepsis and has shown a significant correlation with other relatively expensive and non-rapidly existing markers of inflammation and sepsis.

Importantly, research on NLR in sepsis has received wide attention in recent years. NLR within 24 hours before intensive care unit (ICU) admission could be used as a marker for early diagnosis of sepsis. In addition to the diagnostic value of NLR, it is worth mentioning that NLR has also been found to have the ability of predicting the prognosis of sepsis. A meta-analysis in 2019 indicates that peripheral blood leucocyte ratios, including NLR, lymphocyte-to-monocyte ratio (LMR) and platelet-to-lymphocyte ratios (PLR), could be useful infection biomarkers and associated with clinical prognosis of sepsis. A meta-analysis in 2020 also indicates that the higher NLR was linked to poor prognosis in patients with sepsis (n = 10,685) (hazard ratio (HR) = 1.75). NLR at admission is shown to be an independent predictor of in-hospital mortality of septic patients (n = 174). NLR, PLR and LMR can be useful predictors for early identification of post-percutaneous nephrolithotomy (PNL) sepsis. However, the exact role of NLR in the early prediction of the prognosis of septic patients remain controversial. No correlation was found between NLR at admission of emergency department and 28-day hospital mortality of septic patients. NLR at admission is less suitable than conventional inflammatory markers C-reactive protein (CRP) and procalcitonin (PCT) to detect the presence of sepsis in ICU patients. NLR at ICU admission is also less reliable than CRP, PCT, lactic acid and acute physiology and chronic health evaluation (APACHE Ⅱ) score in assessing the severity and in predicting 28-day mortality of critical illness.

In this study, the investigators enrolled septic patients to determine the role of NLR in the early prediction of in-hospital mortality of patients with sepsis. In addition, considering that PLR, neutrophil percentage (NE%) and monocyte to lymphocyte ratio (MLR) have been confirmed to be also associated with the mortality of patients with sepsis, while retrospectively analyzing the role of NLR, the investigators also studied the roles of PLR, MLR, neutrophil percentage, and other inflammation-related parameters on the first, second, third, and seventh days after hospitilization in the in-hospital mortality of septic patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with sepsis
* 2.ICU stay time ≥3 days;

Exclusion Criteria:

* 1. History of solid organ or bone marrow transplantation;
* 2. Diseases that may affect immune-related indicators, such as autoimmune diseases such as rheumatoid arthritis and SLE, or hematological malignancies such as leukemia and lymphoma;
* 3. Have received radiotherapy or chemotherapy within the past 30 days, or have received immunosuppressive drugs (tripterygium, mycophenolate, cyclophosphamide, FK506, etc.), or have received continuous treatment with more than 10mg of prednisolone/day (or the same dose of other hormones);
* 4. Pregnancy or lactation;c

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed sepsisc
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
NLR | day 1, day2, day 3, and day 7 after admission.
  NLR values were collected on day 1, day 2, day 3, and day 7 after admission.

SECONDARY OUTCOMES:
NE% | on day 1, day 2, day 3, and day 7 after admission.
  NE% were collected on day 1, day 2, day 3, and day 7 after admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang M, Cai S, Su J. The Pathogenesis of Sepsis and Potential Therapeutic Targets. Int J Mol Sci. 2019 Oct 29;20(21):5376. doi: 10.3390/ijms20215376. PMID 31671729
- [Background] Ji J, Fan J. Neutrophil in Reverse Migration: Role in Sepsis. Front Immunol. 2021 Mar 15;12:656039. doi: 10.3389/fimmu.2021.656039. eCollection 2021. PMID 33790916
- [Background] Manz MG, Boettcher S. Emergency granulopoiesis. Nat Rev Immunol. 2014 May;14(5):302-14. doi: 10.1038/nri3660. Epub 2014 Apr 22. PMID 24751955
- [Background] Grailer JJ, Fattahi F, Dick RS, Zetoune FS, Ward PA. Cutting edge: critical role for C5aRs in the development of septic lymphopenia in mice. J Immunol. 2015 Feb 1;194(3):868-72. doi: 10.4049/jimmunol.1401193. Epub 2014 Dec 24. PMID 25539817
- [Background] Zahorec R. Neutrophil-to-lymphocyte ratio, past, present and future perspectives. Bratisl Lek Listy. 2021;122(7):474-488. doi: 10.4149/BLL_2021_078. PMID 34161115
- [Background] Rehman FU, Khan A, Aziz A, Iqbal M, Mahmood SBZ, Ali N. Neutrophils to Lymphocyte Ratio: Earliest and Efficacious Markers of Sepsis. Cureus. 2020 Oct 8;12(10):e10851. doi: 10.7759/cureus.10851. PMID 33178505
- [Background] Martins EC, Silveira LDF, Viegas K, Beck AD, Fioravantti Junior G, Cremonese RV, Lora PS. Neutrophil-lymphocyte ratio in the early diagnosis of sepsis in an intensive care unit: a case-control study. Rev Bras Ter Intensiva. 2019;31(1):64-70. doi: 10.5935/0103-507X.20190010. Epub 2019 Mar 21. PMID 30916236
- [Background] Ni J, Wang H, Li Y, Shu Y, Liu Y. Neutrophil to lymphocyte ratio (NLR) as a prognostic marker for in-hospital mortality of patients with sepsis: A secondary analysis based on a single-center, retrospective, cohort study. Medicine (Baltimore). 2019 Nov;98(46):e18029. doi: 10.1097/MD.0000000000018029. PMID 31725679
- [Background] Russell CD, Parajuli A, Gale HJ, Bulteel NS, Schuetz P, de Jager CPC, Loonen AJM, Merekoulias GI, Baillie JK. The utility of peripheral blood leucocyte ratios as biomarkers in infectious diseases: A systematic review and meta-analysis. J Infect. 2019 May;78(5):339-348. doi: 10.1016/j.jinf.2019.02.006. Epub 2019 Feb 22. PMID 30802469
- [Background] Huang Z, Fu Z, Huang W, Huang K. Prognostic value of neutrophil-to-lymphocyte ratio in sepsis: A meta-analysis. Am J Emerg Med. 2020 Mar;38(3):641-647. doi: 10.1016/j.ajem.2019.10.023. Epub 2019 Nov 18. PMID 31785981
- [Background] Kriplani A, Pandit S, Chawla A, de la Rosette JJMCH, Laguna P, Jayadeva Reddy S, Somani BK. Neutrophil-lymphocyte ratio (NLR), platelet-lymphocyte ratio (PLR) and lymphocyte-monocyte ratio (LMR) in predicting systemic inflammatory response syndrome (SIRS) and sepsis after percutaneous nephrolithotomy (PNL). Urolithiasis. 2022 Jun;50(3):341-348. doi: 10.1007/s00240-022-01319-0. Epub 2022 Mar 4. PMID 35246692
- [Background] Liu Y, Zheng J, Zhang D, Jing L. Neutrophil-lymphocyte ratio and plasma lactate predict 28-day mortality in patients with sepsis. J Clin Lab Anal. 2019 Sep;33(7):e22942. doi: 10.1002/jcla.22942. Epub 2019 Jul 2. PMID 31265174
- [Background] Chebl RB, Assaf M, Kattouf N, Haidar S, Khamis M, Abdeldaem K, Makki M, Tamim H, Dagher GA. The association between the neutrophil to lymphocyte ratio and in-hospital mortality among sepsis patients: A prospective study. Medicine (Baltimore). 2022 Jul 29;101(30):e29343. doi: 10.1097/MD.0000000000029343. PMID 35905272
- [Background] Westerdijk K, Simons KS, Zegers M, Wever PC, Pickkers P, de Jager CPC. The value of the neutrophil-lymphocyte count ratio in the diagnosis of sepsis in patients admitted to the Intensive Care Unit: A retrospective cohort study. PLoS One. 2019 Feb 27;14(2):e0212861. doi: 10.1371/journal.pone.0212861. eCollection 2019. PMID 30811475
- [Background] Zhou T, Zheng N, Li X, Zhu D, Han Y. Prognostic value of neutrophil- lymphocyte count ratio (NLCR) among adult ICU patients in comparison to APACHE II score and conventional inflammatory markers: a multi center retrospective cohort study. BMC Emerg Med. 2021 Feb 23;21(1):24. doi: 10.1186/s12873-021-00418-2. PMID 33622247
- [Background] Can E, Hamilcikan S, Can C. The Value of Neutrophil to Lymphocyte Ratio and Platelet to Lymphocyte Ratio for Detecting Early-onset Neonatal Sepsis. J Pediatr Hematol Oncol. 2018 May;40(4):e229-e232. doi: 10.1097/MPH.0000000000001059. PMID 29219889
- [Background] Tian T, Wei B, Wang J. Study of C-reactive protein, procalcitonin, and immunocyte ratios in 194 patients with sepsis. BMC Emerg Med. 2021 Jul 7;21(1):81. doi: 10.1186/s12873-021-00477-5. PMID 34233608
- [Background] Meshaal MS, Nagi A, Eldamaty A, Elnaggar W, Gaber M, Rizk H. Neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR) as independent predictors of outcome in infective endocarditis (IE). Egypt Heart J. 2019 Sep 18;71(1):13. doi: 10.1186/s43044-019-0014-2. PMID 31659520